CLINICAL TRIAL: NCT04774107
Title: An Open-label Study to Assess the Pharmacokinetics of P1101 + Ribavirin in Interferon Treatment-Naïve Subjects With Chronic Hepatitis With HCV Genotype 2 Infection
Brief Title: The Pharmacokinetics of P1101 + Ribavirin in Interferon Treatment-Naïve Subjects With Chronic Hepatitis C Virus (HCV) Genotype 2 Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A20-102
Record Dates: First submitted 2021-01-21; First posted 2021-03-01 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Hepatitis C, Chronic
Keywords: P1101; HCV genotype 2; Pharmacokinetics; PK; Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- P1101 + Ribavirin (Experimental): P1101 400 µg SC Ribavirin 800-1400 mg PO
  Interventions: Drug: P1101 + Ribavirin

INTERVENTIONS:
Drug: P1101 + Ribavirin — P1101 400 µg SC
  Other Names: Ropeginterferon alfa-2b

SUMMARY:
Primary Objective:

To determine the P1101 pharmacokinetic (PK) profile at the single dose of 400 μg.

DETAILED DESCRIPTION:
Secondary Objective:

To determine the safety and immunogenicity of P1101 400 μg subcutaneous (SC) single dose + Ribavirin 800-1400 mg PO daily.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age (or other age required by local regulations); subjects who are over 70 years of age must be in generally good health.
2. Confirmed diagnosis of chronic hepatitis with HCV genotype 2 infection.
3. Compensated liver disease defined by normal or elevated alanine transaminase (ALT) ≤10 x upper limit of normal (ULN), total bilirubin level <2 mg/dL (except in Gilbert's syndrome), normal albumin, normal international normalized ratio (INR)
4. Interferon treatment naïve: never received any interferon.
5. No other known form of chronic liver disease apart from chronic hepatitis C infection.
6. Hemoglobin 12 g/dL in men or 11 g/dL in women, white blood cell (WBC) count 3,000/mm3, absolute neutrophil count (ANC) 1,500/mm3, platelet count 90,000/mm3; and estimated glomerular filtration rate >60 mL/min.
7. Female and male subjects, and their partners of reproductive potential using effective means of contraception during the whole trial period.
8. Be able to attend all scheduled visits and to comply with all study procedures;
9. Be able to provide written informed consent.

Exclusion Criteria:

1. Decompensated liver disease.
2. Clinically significant illness or surgery within 4 weeks prior to dosing.
3. Any reason which, in the opinion of the investigator, would prevent the subject from participating in the study.
4. Positive test for HBsAg or HIV at screening.
5. Clinically significant abnormal vital signs.
6. Evidence of severe retinopathy by fundoscopy except age-related macular degeneration.
7. Significant alcohol or illicit drug abuse within one year prior to the screening visit or refusal to abstain from excessive alcohol consumption as defined above or illicit drugs throughout the study.
8. Pregnant or breast feeding female subjects.
9. Therapy with any systemic anti-viral, anti-neoplastic, and immunomodulatory treatment.
10. Use of an investigational drug or participation in an investigational drug.
11. Known clinically significant presence of any gastrointestinal pathology, clinically significant unresolved gastrointestinal symptoms, clinically significant liver or clinically significant kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
12. Clinically significant presence of depression determined by investigators.
13. Clinically significant presence of severe neurological disorders.
14. Clinically significant presence of severe cardiovascular conditions and severe pulmonary conditions, uncontrolled immunologic, uncontrolled autoimmune, uncontrolled endocrine, uncontrolled metabolic, haematological, severe coagulation disorders or severe blood dyscrasias or other severe uncontrolled systemic disease.
15. A depot injection or an implant of any drug within 3 months prior to administration of study medication, other than contraception or hyaluronic acid injections in joints for osteoarthritis;
16. Body organ transplant and are taking immunosuppressants;
17. History of malignant disease, including solid tumors and hematologic malignancies. However, subjects who are cancer survivors not on maintenance therapy and who had no malignant diseases history within the past 5 years could be recruited.
18. History of or ongoing opportunistic infection.
19. Serious local infection or systemic infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Amount of P1101 in the blood stream | 2-4 weeks
  The measurement of P1101 levels in the blood stream over time. The sampling time points are 0 hour before the first dose, 24±4 hours, 48±4 hours, 72±4 hours, 96±4 hours, 168±4 hours, 216±4 hours, 264±4 hours and 336±4 hours after first dose. PK sampling at 504±4 hours and 672±4 hours after first dose are optional.

SECONDARY OUTCOMES:
Adverse Events | 2-4 weeks
  To evaluate the safety of P1101 by the proportion of adverse events
Abnormal Laboratory Assessments | 2-4 weeks
  To evaluate the safety of P1101 by the proportion of abnormal laboratory assessments
Positive anti-drug antibodies | 2-4 weeks
  To evaluate the positive anti-drug antibodies of P1101 by the proportion
Positive neutralizing antibody | 2-4 weeks
  To evaluate the positive neutralizing antibody of P1101 by the proportion

CONTACTS AND LOCATIONS:
Overall Officials: Huang Yi-Wen, MD/PhD, Study Director — PharmaEssentia
Locations (5):
- Taiwan (5):
  - Chang Gung Memorial Hospital, Chiayi Branch, Chiayi City
  - Chia-Yi Christian Hospital, Chiayi City
  - St. Martin De Porres Hospital, Chiayi City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chi Mei Medical Center, Tainan